CLINICAL TRIAL: NCT02323529
Title: Open-label, Multicentre, Multiple-dose Trial to Evaluate Pharmacokinetics, Efficacy and Safety of Once Daily Dosing Compared to Twice Daily Dosing of Orfadin in Patients Diagnosed With Hereditary Tyrosinemia Type 1
Brief Title: Efficacy and Safety of Once Daily Dosing Compared to Twice Daily Dosing of Nitisinone in HT-1
Acronym: HT-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Sobi.NTBC-003
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Hereditary Tyrosinemia, Type I
Keywords: Orfadin; Nitisinone; NTBC
MeSH Terms: conditions — Tyrosinemias | interventions — nitisinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nitisinone treatment group (Experimental): All patients in the study will first be put on twice daily dosing of nitisinone for 4 weeks. This will then be followed by once daily dosing of nitisinone for 4 weeks.
  Interventions: Drug: Nitisinone

INTERVENTIONS:
Drug: Nitisinone — All patients in the study will first be put on twice daily dosing of nitisinone for 4 weeks. This will then be followed by once daily dosing of nitisinone for 4 weeks. The dose of nitisinone in the study will be the same as the one prescribed at completed screening visit. Dose will be 1-2 mg/kg body weight.
  Other Names: Orfadin

SUMMARY:
The purpose of this study is to look at the steady-state serum concentrations of nitisinone when switching from twice daily and once daily dosing.

DETAILED DESCRIPTION:
Nitisinone (Orfadin) is used in the treatment of hereditary tyrosinemia type 1(HT-1), an inborn error of metabolism. The clinical study that forms the basis for licensing of nitisinone in the treatment of HT-1 used twice daily dosing. This became the recommended dosing frequency of nitisinone stated in the Summary of Product Characteristics. Later on, when the half-life became know (around 50 hours in adults), many physicians started to use once daily dosing. The suitability of once daily dosing and especially of switching patients from twice to once daily dosing has not been documented. The aim with this study is therefore to investigate the effect on nitisinone serum concentrations (Cmax and Cmin) and possible clinical consequences of a lower dosing frequency.

This one-way crossover study consists of three periods; Screening period, Treatment period 1 and Treatment period 2. The study starts with a screening period (Visit 1-1b) that may be up to 6 weeks long. This is followed by two treatment periods of at least 4 weeks each. During Treatment period 1 (Visits 2-3), the patient will take Orfadin twice daily. During Treatment period 2 (Visits 4-5), the patient will take Orfadin once daily. The dose of nitisinone in the study will be the same as the one prescribed at completed screening visit. Dose will be 1-2 mg/kg body weight. The total treatment period will be at least 8 weeks.

At least 20 patients with a minimum of 3 patients in each of the following age groups will be included; infants (< 2 years), children (2-<12 years), adolescents (12-<18 years) and adults (≥18 years).

Determination of succinylacetone (SA) in blood (serum/plasma) and/or urine will be performed both locally and at a central Good Laboratory Practice certified laboratory (Dry Blood Spot sample). The purpose of the local sample is to provide the investigator with more or less immediate results to determine if a dose adjustment is needed before the patient enters either of the two treatment periods. Results from samples analyzed at the central laboratory, including determination of nitisinone, will be used in the evaluation of pharmacokinetics, efficacy and safety during the two treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of all ages diagnosed with HT-1.
* Patients currently well-controlled, as judged by the investigator, on twice daily (or more frequent) dosing with Orfadin.
* Stable lab values, including liver values <2 ULN (ALP, ALT, AST, bilirubin, INR).
* Women of childbearing potential willing to use adequate contraception
* Signed informed consent/assent.

Exclusion Criteria:

* Patients who have been previously treated with once daily Orfadin, even if later converted to twice daily dosing.
* Any medical condition which in the opinion of the investigator makes the patient unsuitable for inclusion.
* Enrollment in another concurrent clinical interventional study within three months prior to inclusion in this study.
* Pregnant women.
* Lactating women.
* Previous liver transplantation.
* Patients who have recently (past 4 weeks prior to inclusion) started any new medication for a previously undiagnosed illness/disease.
* Known hepatitis B, hepatitis C or HIV infection.
* Foreseeable inability to cooperate with given instructions or study procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Minimum serum concentration (Cmin) of nitisinone | 4 weeks
  Sample collected immediately before administration of morning dose

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) of nitisinone | 4 weeks
  Sample collected 3-4 hours post dose
Cmax/Cmin ratio of nitisinone | 4 weeks
Number of patients with Serum succinylacetone (s-SA) above lower limit of quantification (LLOQ) | 4 weeks
Minimum serum concentration (Cmin) of nitisinone at possible occurence of s-SA above lower limit of quantification (LLOQ) | 4 weeks
  Cmin of nitisinone will be listed for patients with s-SA above LLOQ
Number of patients with at least one adverse event | 4 weeks
  Total and by system organ class and preferred term (MedDRA)
Number of patients with at least one serious adverse events | 4 weeks
  Total and by system organ class and preferred term (MedDRA)
Number of patients with at least one study drug related adverse events | 4 weeks
  Total and by system organ class and preferred term (MedDRA)
Number of patients with at least one non-serious adverse event | 4 weeks
  Total and by system organ class and preferred term (MedDRA)
Number of patients with at least one adverse event leading to study discontinuation | 4 weeks
  Total and by system organ class and preferred term (MedDRA)
Serum-tyrosine (µmol/L) | 4 weeks
  Descriptive statistics of s-tyrosine
Serum-alpha fetoprotein (µg/L) | 4 weeks
  Descriptive statistics of s-alpha fetoprotein

CONTACTS AND LOCATIONS:
Overall Officials: Anders Bröijersén, MD, Study Director — Swedish Orphan Biovitrum
Locations (6):
- Swedish Orphan Biovitrum Investigational Site, Brussels, Belgium
- Swedish Orphan Biovitrum Investigational Site, Copenhagen, Denmark
- Swedish Orphan Biovitrum Investigational Site, Lyon, France
- Germany (2):
  - Swedish Orphan Biovitrum Investigational Site, Giessen
  - Swedish Orphan Biovitrum Investigational Site, Reutlingen
- Swedish Orphan Biovitrum Investigational site, Gothenburg, Sweden